CLINICAL TRIAL: NCT06057974
Title: Effects of the Close Collaboration with Parents Intervention on Parents of Newborns
Brief Title: Close Collaboration and Discharge Readiness
Status: Recruiting | Type: Observational
Sponsor: Nagano Children's Hospital (Other)
Responsible Party: Principal Investigator, Ryo Itoshima, Chief physician, Nagano Children's Hospital
Other Study IDs: S-05-49
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Family Centered Care
Keywords: Staff education; Parental anxiety; Parental discharge readiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-intervention: The patient and their parents who are admitted to the NICU before the NICU starts implementing the intervention.
- Post-intervention: The patient and their parents who are admitted to the NICU after the NICU implements the intervention.
  Interventions: Other: Close Collaboration with Parents

INTERVENTIONS:
Other: Close Collaboration with Parents — The Close Collaboration with Parents intervention is an educational model for healthcare staff working in NICUs. It aims to improve the ability of the members of the NICU healthcare team to I) observe the infants' individual behaviors and needs, II) support parents to take the initiative and share their observations and understanding of their infant's behaviors and to collaboratively plan the infant's care with the healthcare staff, III) understand the individual story of the family regarding parenthood through a dialogue with parents, and IV) involve parents in the decision-making about the care of their baby from an early stage of care through to the preparation for discharge. The final goal is to improve the care culture in the NICUs by changing the attitudes of the healthcare staff and the care practices of the unit to be more in line with family-centered care principles.
  It usually takes 1.5 years for each NICU to complete the intervention.
  Groups: Post-intervention

SUMMARY:
This prospective non-randomized controlled before-after comparison study aims to evaluate the effects of the Close Collaboration with Parents, a family-centered care intervention for NICU staff, on parents of the newborns in the neonatal intensive care unit (NICU). We focus on (1) family centered care of the NICU rated by parents, (2) parental anxiety symptoms, and (3) their discharge readiness.

The intervention is planned to be implemented between December 2023 and December 2024.

The investigators will collect data from parents whose newborns are admitted to the NICU before and after the intervention and compare the two groups. In most cases, the parents of the two groups belong to different cohorts.

DETAILED DESCRIPTION:
Study period Pre-intervention data collection phase: September 2023 - December 2023 (Planned) Intervention phase: January 2024 - December 2024 (Planned) Post-intervention data collection phase: January 2025 - April 2025 (Planned)

Outcome measures Primary outcome: Quality of family centered care rated by parents Secondary outcomes: Parental anxiety symptoms and parental discharge readiness

Data management Eligible infants and their information will be identified and collected by research team members and entered into the excel file (.xlsx). Data will be pseudonymized when the data is entered into the excel file. All electronic data will be destroyed 10 years after the initiation of the study.

The principal investigator will be responsible for managing access to the data. We do not have a plan to make the data open in the future.

Statistical analysis The comparison between two continuous variables will be carried out by the student t test and, additionally, the multiple linear regression model and the logistic regression model to adjust the effect of the potential confounders. The potential confounders included in the models will be the length of stay and parents' previous mental illness.

R and RStudio will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Infants who have been admitted to the NICU for 2 weeks or longer

Exclusion Criteria:

* Infants whose parent doesn't have Japanese as their mother tongue
* Infants whose parent needs psychiatric consultation after birth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants and their parents who need at least 2 weeks of admission to Nagano Children's Hospital NICU, a level IV NICU in Japan.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of family centered care rated by parents | at discharge (about 1 month of age)
  The family centered care provided by the medical professionals in the NICU is assessed by parents using a questionnaire modified from DigiFCC questions. It consists of 9 questions. Each question has the Likert scale from 1 to 7 (1 not at all and 7 very much; 0 not applicable). A higher score indicates better family centered care received by parents. The average score of all questions will be used.
  This is rated by both parents separately.

SECONDARY OUTCOMES:
Parental anxiety symptoms | at discharge (about 1 month of age)
  Parents' anxiety is assessed using the short version of the State and Trait Anxiety Inventory (Short-STAI). It was developed based on the original STAI which has 40 questions.9 The STAI assesses two different anxiety types at the same time. State anxiety is an emotional response that can change over time according to the situation. Trait anxiety indicates a personal emotional characteristic that a person has. There are 5 questions for each state and trait anxiety and each is scored on a four-point scale (1-4). The total score in each type of anxiety varies from a minimum of 5 to a maximum of 20, and higher scores indicate having more depressive symptoms.
  This is rated by both parents separately.
Parental discharge readiness | at discharge (about 1 month of age)
  The readiness for the discharge is measured with the Readiness for Hospital Discharge Scale (RHDS). The questionnaire includes 23 items. Four attributes of readiness for discharge are measured within the subscales: Personal Status (7 items), Knowledge (7 items), Coping Ability (4 items), and Expected Support (5 items). Answers are on a 10-point scale from 0 to 10 (e.g., not at all, totally). The RHDS has been shown to be a reliable and valid measure of patients' perception of readiness for discharge. We use Japanese version, whose validity and reliability have also been shown.

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Itoshima, MD, Principal Investigator — Nagano Children's Hospital
Locations (1):
- Nagano Children's Hospita, Azumino, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No